CLINICAL TRIAL: NCT00158093
Title: A Randomized, Parallel Group Safety Evaluation of Electrocardiographic Intervals and Blood Pressure in Normal Healthy Volunteers After Nebivolol, Atenolol, Moxifloxacin, or Placebo Administration After Single and Repeated Doses
Brief Title: A Safety Evaluation of ECG Intervals and Blood Pressure in Normal Healthy Volunteers After Use of Nebivolol, Atenolol, Moxifloxacin, or Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Bertek Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEB122
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Atenolol; Moxifloxacin

INTERVENTIONS:
Drug: Nebivolol
Drug: Atenolol
Drug: Moxifloxacin

SUMMARY:
Nebivolol is one of a class of drugs known as beta-blockers. These drugs are useful in the treatment of high blood pressure, angina, abnormal heart rhythms and following a heart attack. The purpose of this study is to explore the potential of nebivolol to cause a certain type of abnormal heart rhythm, known as QTc prolongation. The potential of nebivolol to cause this adverse event will be compared to three other drugs: atenolol, a beta-blocker approved by the FDA; Avelox (moxifloxacin), an anti-biotic approved for use by the FDA which is known to cause QTc prolongation; and placebo, a drug look-alike that contains no drug. The working hypothesis was that 20 or 40 mg of nebivolol would not prolong corrected QT intervals measured during peak nebivolol concentrations (i.e., 2 hours after dosing) on Day 7.

ELIGIBILITY:
Inclusion Criteria:

* Men and nonpregnant, nonlactating women were 18 years or older.
* Women declaring postmenopausal or surgical sterility.
* Women of childbearing potential who had a negative serum HCG within 2 weeks of dosing.
* Male subjects weighed at least 60 kg (132 lb), and female subjects weighed at least 48 kg (106 lb). All volunteers weighed within 15% of their ideal body weight (IBW).

Exclusion Criteria:

* Institutionalized
* Reported or was known to have done the following:

  * Used any tobacco product.
  * Ingested any alcoholic, caffeine or xanthine containing food or beverage within the 48 hours prior to the initial dose of study medication
  * Consumed grapefruit or grapefruit containing products within 7 days prior to the initial dose of study medication.
  * Ingested any vitamins or herbal products within the 48 hours prior to the initial dose of study medication.
  * Recently changed dietary or exercise habits significantly
* Used any medication (including over-the-counter [OTC]) within the 14 days prior to the initial dose of study medication.
* Used any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
* Received an investigational drug within 30 days prior to the initial dose of study medication.
* History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, or neurologic disease.
* History of drug and/or alcohol abuse within 1 year prior to the study.
* Acute illness at the time of either the pre study medical evaluation or dosing.
* Any laboratory results deemed clinically significant by the physician.
* Abnormal and clinically relevant ECG tracing.
* Donated or lost a significant volume of blood or plasma (>450 mL) within 28 days prior to the initial dose of study medication.
* Allergic or hypersensitive to nebivolol, atenolol, or other β blocking drugs or to moxifloxacin or other quinolone antibiotics.
* History of seizures or cerebrovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260
Dates: Start 2003-06; Study Completion 2003-07

PRIMARY OUTCOMES:
The primary study endpoint was the change in the average QTc intervals from Day 0 to 2 hours after dosing on Day 7.

SECONDARY OUTCOMES:
The secondary endpoints were the change in average QTc intervals from Day 0 to all other evaluation times and the change in other ECG intervals (PR, RR, QRS, QT) and HR from Day 0 to all other evaluation times.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Galitz, MD, Principal Investigator — SFBC International; Will A Sullivan, BS, Study Director — Mylan Bertek Pharmaceuticals Inc.
Locations (1):
- SFBC International, Inc., Miami, Florida, United States